CLINICAL TRIAL: NCT03599492
Title: The Effect of Transjugular Intraheptic Portosystemic Shunt (TIPS) on Gastrointestinal Motility and the Gut Microbiota
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 16-01360
Record Dates: First submitted 2018-07-12; First posted 2018-07-26 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Cirrhosis
Keywords: Gut Microflora; Transjugular Intraheptic Portosystemic Shunting
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cirrhosis Patients: 10 Patients with body mass index (BMI) etiology of cirrhosis
  Interventions: Diagnostic Test: SMART Pill Pre-TIPS; Diagnostic Test: SMART Pill Post TIPS

INTERVENTIONS:
Diagnostic Test: SMART Pill Pre-TIPS — Assessment of motility with Smart Pill, which will be read and confirmed by gastroenterologist trained to interpret motility studies
Diagnostic Test: SMART Pill Post TIPS — Assessment of motility with Smart Pill, which will be read and confirmed by gastroenterologist trained to interpret motility studies

SUMMARY:
The effect of portal hypertension on gastrointestinal motility, and how reversal or improvement in portal hypertension may alter gastrointestinal motility, remains unclear and further research is needed. Additionally, patients with cirrhosis have altered gut microflora, particularly rich in lactobacilli, including enterococci and bifidobacteria. Transjugular Intraheptic Portosystemic Shunting (TIPS) is a procedure performed by interventional radiologists, in which a connection is made between the portal and venous circulations, allowing high pressure portal blood to more easily enter the systemic circulation and bypass the liver; thus effectively decreased portal pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with either radiographic or biopsy proven decompensated cirrhosis (as determined by ascites, variceal hemorrhage, encephalopathy or jaundice).
* Patients undergoing an elective TIPS for any standard of care established indication (examples: worsening ascites, recurrent variceal bleeding).

Exclusion Criteria:

* Pregnant women.
* Patients unwilling or unable to provide informed consent.
* Patients undergoing an emergent TIPS for acute or subacute variceal hemorrhage.
* Patients with diabetes, significant cardiovascular, renal or other chronic disease which has been known to affect intestinal motility.
* Previously diagnosed gastroparesis or other GI dysmotility disorder.
* Patients currently taking narcotics, antibiotics excluding rifaximin, prokinetic medications or lactulose.
* Patients with a history of gastric bezoar.
* Patients with a history of multiple intestinal surgeries or GI surgery within the past 3 months.
* Patients with a history of gastrointestinal strictures, fistulas, or physiological or mechanical obstruction.
* Patients with a history of gastrointestinal strictures, fistulas, or physiological or mechanical obstruction.
* Patients with a history of gastrointestinal strictures, fistulas, or physiological or mechanical obstruction.
* Patients with a history of diverticulitis.
* Patients with swallowing disorders and increased risk of aspiration (such as prior history of aspiration).
* Patient with Celiac disease.
* Patients with implanted or portable electro-mechanical medical devices.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 patients recruited from NYU Langone Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-04-12 (Actual)

PRIMARY OUTCOMES:
Pre-TIPS intestinal transit time (measured in hours and minutes), via smart pill in patients with cirrhosis | 14 Weeks
  Due to small sample size, Wilcoxon rank-sum test will be used to compare the continuous variable of gut transit times. A p-value of <0.05 will be considered statistically significant.
Post TIPS intestinal transit time (measured in hours and minutes), via smart pill in patients with cirrhosis | 14 Weeks
  Due to small sample size, Wilcoxon rank-sum test will be used to compare the continuous variable of gut transit times. A p-value of <0.05 will be considered statistically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Bedros Taslakian, MD, EBIR, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.